CLINICAL TRIAL: NCT05089799
Title: " Socially Pertinent Robot in Gerontological Healthcare "
Acronym: Spring
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other); Università degli Studi di Trento (Other); Czech Technical University in Prague (Other); Heriot-Watt University (Other); ERM Automatismes Industriels (ERM) (Unknown); Pal Robotics SL (PAL) (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201352
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Patient Participation; Patient Relations, Nurse; Professional Role
Keywords: Socially Assistive Robots; Gerontological Healthcare; acceptance; usability; organizational and ethic impact
MeSH Terms: conditions — Patient Participation | interventions — Drug Interactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients: Older adults 60 years old or older They are referred to the day care hospital for memory problems or frailty and may present with various cognitive, behavioural, mental and physical disorders.
  Persons in this group are diverse in socio-cultural levels. The investigators expect to include 100 patients (N = 100). Each patient will test 1 out of the 5 use cases, so 20 patients will test the same use case (n = 20).
  Interventions: Behavioral: Exposure and interaction with a socially assistive robot
- Informal carers or family caregivers: This group includes persons who accompany patients during the hospital visit, such as family members (spouses or children) and friends.
  They provide support to the patient with various frequency and intensity (occasional / regular / continuous).
  Persons in this group are diverse in age and socio-cultural levels. They may also suffer from physical and/or psychological disorders.
  The investigators expect to include 100 informal or family caregivers (N = 100). Each one will test 1 out of the 5 use cases, so 20 informal or family caregivers will test the same use case (n= 20).
  Interventions: Behavioral: Exposure and interaction with a socially assistive robot
- Professionals: All categories of professionals working in the day care hospital. Persons in this group belong to different professional categories (administrative, health, technical). They have different levels of proximity with the public and have various positions in the hospital.
  The investigators expect to include 50 professionals.
  Interventions: Behavioral: Exposure and interaction with a socially assistive robot

INTERVENTIONS:
Behavioral: Exposure and interaction with a socially assistive robot — Description of scenarios involving robot and users
  1. welcoming patients and family members l: the robot explains its own functionalities and answers persons 'questions.
  2. providing a reminder about sanitary gestures (prevention of virus transmission). In addition, it could mediate a conversation between two or more people so that they keep the appropriate physical distance between them.
  3. providing patients with an assistance to prepare the medical consultations : the robot helps patients to fill in paper forms for professionals. The robot also provides information on the course of consultations and the users 'rights in the hospital.
  4. providing orientation and guidance to the consultation rooms and the available services : the robot helps people to find their way around the hospital.
  5. Providing entertainment to patients and families during the waiting time: the robot offers activities to patients and caregivers

SUMMARY:
The SPRING project intends to develop a social assistance robot, called ARI, capable of interacting with several users (patients, families) in noisy and busy hospital environments to inform, guide and entertain them and to support care workers in these environments. The AP-HP researchers participating in the SPRING project wish to evaluate human-robot interactions in a day care hospital and in particular the acceptability and the uses of the robot.

DETAILED DESCRIPTION:
Elderly people suffering from neurocognitive disorders require multimodal support (social, medical, associative) in which Socially Assistive Robots (SARs) could intervene in order to improve the physical and psychological well-being of elderly people and maintain their quality of life. SARs are social entities capable of interacting with their users in a variety of contexts (informational, recreational, educational). These robots also offer promising possibilities for accompanying care workers in their support of people with neurodegenerative diseases. However, up to date, these robots are not sufficiently sophisticated to engage in satisfactory social interactions with human beings and lead to their adoption.

The SPRING study is a non-interventional study that does not include objectives for improving health or patient care. It is an exploratory study targeting five use cases with a social robot and three populations of care hospital users (patients, informal or family caregivers and professionals). No follow-up of the participants is necessary.

The main objective of SPRING is to study the acceptability of socially assistive robots among three actors in a hospital service: patients, informal or family caregivers and professionals. The secondary objectives are to study a) the usability of the ARI robot among day care hospital's users which is necessary to understand the efficiency of using the robot in this context; b) the organisational impact of the robot on the operation of the service among day care hospital's professionals ; c) the ethical questions generated by the presence of the robot with the participants that will allow us to extend our understanding of the determinants of the rejection or adoption of new technologies in the hospital context.

During this non-interventional and exploratory research, the ARI robot will be tested in the waiting room of a day care hospital in a geriatric hospital regarding five use cases (1/welcoming patients and family members to the hospital, 2/ providing a reminder how to follow sanitary gestures for the prevention of virus transmission, 3/providing patients an assistance to prepare for the medical consultation that will follow during the day, 4/ providing orientation and guidance in relation to the location (hospital) and the services available (toilets, cafeteria, elevators, etc.) and 5/Providing entertainment to patients and families during the waiting time.

Patients and their family caregivers meet the robot only once. They answer questionnaires and participate in semi-structured interviews after interacting with the robot. Evaluations target the acceptability, usability and ethical issues raised by the presence of a robotic agent in support of care teams.

The professionals included in the study meet the robot several times according to their professional obligations (hospital practitioners are not present every day at the day care hospital and can choose when to interact with the robot). They will be invited to participate in two focus groups, one before the introduction of the robot and the other one at the end of the study. At the end of the study, the investigators will offer them to fill in questionnaires and participate in semi-structured interviews. The evaluations proposed to the professionals deal with questions of acceptability, usability, organisational impact of the robot's presence, and ethical issues related to its presence in the day care hospital.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS
* Age 60 and over
* Enough knowledge in French language
* Without distinction of gender, socio-professional categories or ethnic origin
* MMSE > 10
* No symptoms of altered reality (delirium, hallucination, frontal disinhibition, etc.).
* Having expressed his/her non-opposition to his/her participation in the study or to being in the presence of the robot
* If the persons are protected adults under guardianship, the tutor or legal guardian has expressed his/her non-opposition to participate in the study or to be in the presence of the robot for the person concerned.
* ACCOMPANYING PERSONS
* They are all adults who have enough knowledge in French language.
* They are enrolled without distinction of gender, socio-professional categories or ethnic origin
* They have expressed his/her non-opposition to participate in the study
* PROFESSIONALS:
* Age 18 and over.
* Has expressed his/her non-opposition to participate in the study

Exclusion Criteria:

* PATIENTS
* They have expressed, or where applicable, their family, guardian or legal representative, their opposition to participate in the study or their opposition to be in the presence of the robot.
* PAtients benefiying of Medical State Aid (French AME)
* ACCOMPANYING PERSONS They are under 18. They do not have enough knowledge in French language to understand simple instructions. They have expressed their opposition to participate in the study or their opposition to be in the presence of the robot.
* PROFESSIONNALS They have expressed their opposition to participate in the study or their opposition to be in the presence of the robot.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population includes the 3 categories of actors attending the day care hospital: patients, their carers (family or close carers) and professionals. The investigators will consider all the actors who are likely to interact with the ARI social robot, including people who are not formally part of the patients' care pathway, but whose presence is important to their care.
  The individuals included will have various profiles, from a demographic, sociological and clinical point of view. The patients and their carers mainly live in the Paris region.
  Patients mainly consult the day care hospital for memory problems, but are likely to display associated cognitive, behavioural or physical problems.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Acceptability E-Scale (AE-S) | Inclusion visit
  This criterion will be evaluated with patients, informal or family caregivers and professionals, on the basis of the French version of the "Acceptability E-Scale" (AE-S), a six items questionnaire rated with a Likert scale from 1 to 5 (Micoulaud-Franchi et al., 2016). The items have been adapted for a use with a robot.
  On the day of the appointment at the day care hospital for patients and their informal or family caregivers. During the experiment for professionals. One session, approximatively 10 minutes length.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Inclusion visit
  The SUS is a 10 items questionnaire rated with a Likert scale from 1 to 5 (Brooke, 1996). Usability will also be evaluated with observations during interactions between participants and the robot.
  On the day of the appointment at the day care hospital for patients and their carers. During the experiment for professionals. On session, approximatively, 15 minutes length.
Semi-structured interview (10 questions) based on the USUS model (Hebesberger et al., 2017) | Inclusion visit
  The organisational impactwill be evaluated with the professionals at the end of the experiment using a semi-structured interview (10 questions) based on the USUS model (Hebesberger et al., 2017).
  During the experiment for professionals. One session, approximatively 15 minutes length.
Semi-structured interview (6 questions) | Inclusion visit
  Ethical aspects will be assessed by means of a semi-structured interview (6 questions) with day care hospital's users based on the ethical questions included in the acceptability questionnaire based on the UTAUT model (Alaiad & Zhou, 2014) and through an adaptation of some items of the "Ethical Acceptability Scale" (Peca, 2016).
  On the day of the appointment at the day care hospital for patients and their carers. During the experiment for professionals. One session, approximatively 15 minutes length.

CONTACTS AND LOCATIONS:
Overall Officials: RIGAUD Anne-Sophie, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris (AP-HP) - Broca Hospital - Geriatric unit, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
The robot will process audio-visual data, using object, body and face localisation technologies as well as multi-microphone sound localisation to track objects and people and map the dynamics of its environment. The robot will also analyse facial features in order to decipher the emotional states of participants and trigger appropriate behaviour. However, the robot will not perform any profiling as defined by General Data Protection Regulation (GDPR): it will not process the data it collects in order to individualise or categorise a person. Furthermore, the robot's memory will be erased every night.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD collected by the robot will be available from the start of the study and kept for up to two years after the first publications.
Access Criteria: The data collected by the robot will be stored on a server at the AP-HP at BLL and then transmitted to INRIA engineers according to a secure transfer protocol with cryptographic method: End to end encryption (https, SSH, key/certificate authentication). The data will be transmitted to the SPRING project partners according to secure transfer and storage protocols, validated by the INRIA Defence Security Officer, to ensure the best conditions of confidentiality and security.

REFERENCES:
- [Background] Blavette L, Dacunha S, Alameda-Pineda X, Hernandez Garcia D, Gannot S, Gras F, Gunson N, Lemaignan S, Polic M, Tandeitnik P, Tonini F, Rigaud AS, Pino M. Acceptability and Usability of a Socially Assistive Robot Integrated With a Large Language Model for Enhanced Human-Robot Interaction in a Geriatric Care Institution: Mixed Methods Evaluation. JMIR Hum Factors. 2025 Aug 1;12:e76496. doi: 10.2196/76496. PMID 40750072
- See also: The page presents the SPRING project and all the contributors of the project. — http://spring-h2020.eu/